CLINICAL TRIAL: NCT07088276
Title: Microneedling Combined With Topical Crisaborole 2 % Ointment in Treatment of Vitiligo. A Prospective Controlled Trial.
Brief Title: Microneedling Combined With Topical Crisaborole 2 % Ointment in Treatment of Vitiligo.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Hassan Moustafa Fahmy, Lecturer of Dermatology and Venereology, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS976/6/25
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Percutaneous Collagen Induction; crisaborole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the main patch with microneedling and topical crisaborole and two patches as control (Other): each patient will have 3 vitiligo patches one will be treated by microneedling and topical application of crisaborole and the other 2 patches will be considered as control patches
  Interventions: Procedure: microneedling with topical crisaborole

INTERVENTIONS:
Procedure: microneedling with topical crisaborole — From each patient 3 patches will be selected The first will have microneedling and topical crisaborole and NB UVB sessions The second will have microneedling and NB UVB sessions The third will be exposed only to NB UVB sessions The microneedling sessions will be every 2 weeks for 6 sessions

SUMMARY:
The goal of this clinical trial is to learn if topical crisaborole ointment works to treat vitiligo. It will also learn about the safety of the drug. The main questions it aims to answer are:

Can the drug cause repigmentation of vitiligo lesions when used as topical form after microneedling? What medical problems do participants have when the drug used?

Participants will:

Visit the clinic once every 2 weeks to have the microneedling sessions for 3 months. and also they will have narrow band UVB sessions two times per week.

Record any side effect they have during or after the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffer from non-segmental stable vitiligo.
* Patients who will accept to be included in the study and will sign a written consent.

Exclusion Criteria:

* Patients with history of koebnerization or any sign of disease activity.
* Patients with keloid tendency.
* Patients with active infection.
* Pregnant or lactating woman.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Repigmentation of vitiligo lesions | 3 months from the start of treatment
  The repigmentation responses will be expressed qualitatively as the following No change (0%-25%) = mild improvement (26%-50%) = moderate improvement (51%-75%) = good improvement (76%-100%) = excellent improvement